CLINICAL TRIAL: NCT04617184
Title: Registry and Biorepository for the Study of Inflammatory Bowel Diseases in Central Texas
Brief Title: Registry and Biorepository for IBD in Central Texas
Status: Recruiting | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Linda Anne Feagins, MD, Associate Professor of Medicine, University of Texas at Austin
Other Study IDs: 2019-07-0137
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease: any patient with IBD will be included in the registry
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — THERE IS NO INTERVENTION TO THIS TRIAL. THIS IS A REGISTRY

SUMMARY:
This is a prospective, non-interventional registry and biorepository for patients with IBD. Longitudinal follow-up data is collected from both patients and their treating gastroenterologist during routine clinical encounters. The biorepository will consist of prospective collection of blood samples, tissue samples, and fecal samples for research purposes, while the participants are undergoing a clinically-indicated procedure (i.e. venipuncture for routine tests, IV catheter placement, and/or endoscopy). Participants may choose to provide any or all of the aforementioned information and/or samples.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* Willing and able to provide written consent for participation in the registry and biorepository
* Patients with known or suspected inflammatory bowel disease

Exclusion Criteria:

* Patient is unable to comprehend and/or cooperate with study activities
* Patient is too ill to provide consent
* Coagulopathy that precludes safe biopsy of the bowel
* Comorbidity that precludes safe participation in endoscopic procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with a diagnosis or suspected diagnosis of IBD made by the treating medical team will be considered for recruitment and enrollment. No special populations are targeted for accrual to this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with inflammatory bowel disease | 10 YEARS
  Number of patients with Crohns, ulcerative colitis, and IBD undetermined

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Medical School, UT Austin, Austin, Texas, United States